CLINICAL TRIAL: NCT03867552
Title: Pain Relief in Laparoscopic Surgery - to Relief Pain After Laparoscopic Surgery With the Use of a Altered Gas
Brief Title: Pain Relief in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Anesthesiologist, MD, PhD, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19.08/Gynaeco19.01
Record Dates: First submitted 2019-02-28; First posted 2019-03-08 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative; Surgery
Keywords: post-operative pain; recovery; laparoscopy; nitrous oxide
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A total of 4 conditions will be assessed: endometriosis, myoma, hysterectomy and colpopexy. For every group of patients receiving the altered gas, a group of controls which are patients receiving the standardized gas will be assessed to compare the results in a double-blinded fashion
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Altered gas (86% CO2, 10% N2O, 4% O2) (Experimental): Surgery with the use of the altered insufflation gas (86% CO2, 10% N2O, 4% O2)
  Interventions: Procedure: Altered gas (86% CO2, 10% N2O, 4% O2)
- Standard gas (100% CO2) (Active Comparator): Surgery with the use of the standardized gas (100% CO2)
  Interventions: Procedure: Standardized gas (100% CO2)

INTERVENTIONS:
Procedure: Altered gas (86% CO2, 10% N2O, 4% O2) — Assessment of pain degree after laparoscopic surgery with the altered gas (86% CO2, 10% N2O, 4% O2)
  Arms: Altered gas (86% CO2, 10% N2O, 4% O2)
Procedure: Standardized gas (100% CO2) — Assessement of pain degree after laparoscopic surgery with the standardized gas (100% CO2)
  Arms: Standard gas (100% CO2)

SUMMARY:
Pain relief after laparoscopic surgery with the use of an altered gas.

DETAILED DESCRIPTION:
Pain after laparoscopic surgery remains an important concern in the treatment of endometriosis or other gynaecologic laparoscopic surgery. Several trials have demonstrated that the use of an altered insufflation gas (10 % nitrous oxide + 4% oxygen + 86% carbon dioxide) reduces pain. It also decreases inflammation and adhesion formation as a surplus.

With this mono-center, investigator initiated, double-blinded, randomized controlled superiority trial, the investigators want to demonstrate a reduced postoperative pain and peritoneal inflammatory reaction following peritoneal conditioning with an altered insufflation gas compared to the standard carbon dioxide (100% CO2) insufflation gas. Therefore, women undergoing laparoscopic (gynaecological) surgery with an estimated surgical time of >60 minutes will be asked to participate in this trial. Baseline characteristics will be assessed, including the patients' age, body mass index, medial history, American Society of Anesthesiologist Classification (ASA classification), work status, highest level of education, fear for the surgical procedure (using an 8-item surgical fear questionnaire), pre-operative pain (using a Numerical Rating Scale (NRS) were 0= no pain and 10= worst pain imaginable) both in resting position and in an active position), expected pain (NRS), baseline quality of recovery (QOR) (using the 1-item Global Surgical Recovery (GSR) index (3) and the Functional Recovery Index (FRI) (4)) as well as baseline quality of Life (QOL), using the 5-dimensional European Quality of Life (EQ-5D) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years old
* undergoing laparoscopic surgery for endometriosis, uterine myoma's, hysterectomy or colpopexy.

Exclusion Criteria:

* Women < 18 years old
* Males
* Pregnancy
* Conditions associated with chronic pain, such as peripheral neuropathy, pathology of the vertebral column and osteo-articular disease.
* Conditions causing acute pain e.g. abdominal trauma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation
Enrollment: 74 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Assessment of post-operative pain with an 11-point numerical rating score (NRS) | 4 hours after laparoscopic surgery
  Assessement of pain after laparoscopic surgery with the use of the altered gas compared to standard gas with NRS, where 0 means no pain and 10 means worst imaginable pain

SECONDARY OUTCOMES:
Assessment of post-operative pain (NRS) | 8 hours, 24 hours and 7 days after laparoscopic surgery
  Assessement of pain at different time points after surgery with an 11-point numerical rating score NRS, where 0 means no pain and 10 means worst imaginable pain
Nausea | 4 hours, 8 hours, 24 hours and 7 days after laparoscopic surgery
  Assessment of nausea at different time points after surgery (yes/no)
Post-operative use of piritramide (Dipidolor®) | Up to 24 hours after laparoscopic surgery
  Dose of piritramide after laparoscopic surgery in patients treated with altered gas compared to patients treated with the standard gas
Assessment of degree of a possible inflammatory reaction | Through study completion, up to 7 days after laparoscopic surgery
  Assessed via standard medical practice: body temperature will be measured in °C in order to investigate fever
Assessment of degree of a possible inflammatory reaction | Through study completion, up to 7 days after laparoscopic surgery
  Assessed via standard medical practice: potential blood samples measuring C-Reactive Protein (in mg/l) which is a measure for inflammation can be measured if needed throughout the study
Time to resumption of transit | Through study completion, up to 7 days after laparoscopic surgery
  Time to first flatus and time to first stool
Assessment of quality of Recovery (QOR) | 24 hours and 7 days after laparoscopic surgery
  Assessment of QOR using the 1-item Global Surgical Recovery (GSR) index which represents a single question about the extent to which patients considered themselves to be recovered from surgery ("if 100% recovery means the participants health is back to the same level as it was before the surgery, what percentage of recovery is the participant at now")
Assessment of quality of Recovery (QOR) | 24 hours and 7 days after laparoscopic surgery
  Assessment of QOR using the Functional Recovery Index (FRI) questionnaire which assesses functional QOL on an NRS scale and covers 14 items grouped under three factors (pain and social activity, lower limb activity and general physical activity)
Patient satisfaction | 7 days after laparoscopic surgery
  Assessement of patient satisfaction via a seven-point Likert scale, where 1 means extremely unsatisfied and 7 means extremely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Björn Stessel, MD, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided